CLINICAL TRIAL: NCT03909230
Title: Endometrial Fluid Study in Natural Cycles: a Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Anecova SA (Industry)
Responsible Party: Sponsor
Other Study IDs: NCV-VIS-001
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Endometrial Fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Day 2 post ovulation: Ultrasound of the endometrium, Endometrial fluid sample, Blood sample
- Day 4 post ovulation: Ultrasound of the endometrium, Endometrial fluid sample, Blood sample

SUMMARY:
This study is designed to collect information about the characteristics of endometrial fluid at day 2 and day 4 post-ovulation in normal fertile women.

DETAILED DESCRIPTION:
Implantation rates have stabilised around 35% in IVF and a current key rate limiting step is achieving successful implantation of the embryo. 1/3 of implantation failures are estimated to be caused by a problem with the receptivity of the endometrium. In recent years, several measurable parameters have been reported to assess endometrial receptivity. However, one parameter remains undescribed, the endometrial fluid viscosity.

It is generally believed that the viscosity change post ovulation is influenced by the luteal phase endocrine milieu, and it is possible that the viscosity of the endometrial fluid has an impact on implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 35 years
* Women eligible and qualified for egg donation at IVIRMA Bilbao
* Proven fertile (having given birth to at least one spontaneously conceived normal child)
* Signed written consent including sharing of anonymized data

Exclusion Criteria:

* Contraindications for egg donation according to IVIRMA Bilbao guidelines

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women eligible and qualified as egg donors at IVIRMA Bilbao that meets the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Viscosity of endometrial fluid at D2 and D4 post ovulation of the normal cycle, respectively | 4 days

SECONDARY OUTCOMES:
Plasma progesterone level | 4 days
Plasma estradiol (E2) level | 4 days
Endometrial thickness as measured by ultrasound | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- IVIRMA Bilbao, Leioa, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No